CLINICAL TRIAL: NCT03181217
Title: Functional Magnetic Resonance Imaging of Human Hypothalamic Responses to Oral Temperature and Glucose Sensing
Acronym: COLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FDS-BNH-0770
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- water 22, water 0, glucose 0, glucose 22 (Experimental): Subjects consume 300 ml water at 22 ºC, 300 ml water at 0 ºC, 300 ml water at 0 ºC containing 75 grams glucose and 300 ml water at 22 ºC containing 75 grams glucose sequentially with a one-week washout between consumptions
  Interventions: Other: water 0; Other: water 22; Other: Glucose 0; Other: Glucose 22
- water 0, glucose 22, water 22, glucose 0 (Experimental): Subjects consume 300 ml water at 0 ºC, 300 ml water at 22 ºC containing 75 grams glucose, 300 ml water at 22 ºC and 300 ml water at 0 ºC containing 75 grams glucose sequentially with a one-week washout between consumptions
  Interventions: Other: water 0; Other: water 22; Other: Glucose 0; Other: Glucose 22
- glucose 22, glucose 0, water 0, water 22 (Experimental): Subjects consume 300 ml water at 22ºC containing 75 grams glucose, 300 ml water at 0 ºC containing 75 grams glucose, 300 ml water at 0 ºC and 300 ml water at 22 ºC sequentially with a one-week washout between consumptions
  Interventions: Other: water 0; Other: water 22; Other: Glucose 0; Other: Glucose 22
- glucose 0, water 22, glucose 22, water 0 (Experimental): Subjects consume 300 ml water at 0 ºC containing 75 grams glucose, 300 ml water at 22 ºC, 300 ml water at 22 ºC containing 75 grams glucose and 300 ml water at 0 ºC sequentially with a one-week washout between consumptions
  Interventions: Other: water 0; Other: water 22; Other: Glucose 0; Other: Glucose 22

INTERVENTIONS:
Other: water 0 — 300 ml tap water at 0 ºC
Other: water 22 — 300 ml tap water at 22 ºC
Other: Glucose 0 — 300 ml tap water at 0 ºC with 75 grams of glucose added
Other: Glucose 22 — 300 ml tap water at 22 ºC with 75 grams of glucose added

SUMMARY:
The study will consist of four occasions with one week between the occasions. fMRI will be performed to monitor hypothalamic activity before and after an ingestion of 1 of the following 4 stimuli (300 ml of each): water at room temperature, water at 0 degrees Celsius, glucose solution at room temperature, glucose solution at 0 degrees Celsius. The last two stimuli both contain 75 gram glucose. The order of conditions will be randomly assigned to the subjects. Functional connectivity of the hypothalamic regions will be assessed by analysing the resting state fMRI.

DETAILED DESCRIPTION:
Background of the study: Thermo-regulation is an important aspect of human homeostasis. A decrease in brain and/or body temperature will increase energy requirements and eventually food intake, which acts as a defence against hypothermia. The hypothalamus plays a central role in the regulation of temperature as well as in the control of energy intake, feeding behaviour and lipid and glucose metabolism. The effect of both cooling and changes in energy demand, will therefore be reflected in hypothalamic activity.

Functional magnetic resonance imaging (fMRI) is a non-invasive method, which detects transient haemodynamic changes in the brain, using blood oxygen level dependent (BOLD) signal differences in response to external or internal stimuli. Recently, several fMRI studies have shown the feasibility of measuring hypothalamic function in response to glucose ingestion.

In order to investigate the role of hypothalamic neural activity in response to cooling by food temperature and the additional effect of glucose concentration, fMRI will be performed in healthy men after ingestion of one of 4 solutions at different temperatures and with different glucose concentration.

The study will consist of four occasions. There will be an interval of at least one week between the occasions. On all occasions, the subject will be admitted to the Clinical Research Unit of the LUMC. After a acclimatisation period of 30 minutes and anthropometric measurements (weight and height), fMRI to monitor hypothalamic activity will be performed after an ingestion of 1 of the following 4 stimuli (300 ml of each): water at room temperature, water almost frozen (0 C), glucose solution at room temperature, almost frozen glucose solution (0 C). The last two stimuli both contain 75 gram glucose. Conditions will be randomly assigned to the subjects, a batch wise randomisation procedure will be followed. The order of allocation of each subject is recorded on paper and stored in a sealed envelop, which will be opened after inclusion in the study. The hypothalamus will be continuously imaged for 20 min. (8 min baseline, 4 min drinking, 8 min post ingestion) using a conventional T2*-weighted gradient-echo pulse sequence. A resting state fMRI will be carried out before and after the fMRI of the hypothalamic activity. Hedonic changes or reward effects of the administration will be captured by separate analysis of the amygdala and nucleus accumbens in each subject.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 25 years
* BMI between 20 and 23 kg/m2
* Length between 170 and 190 centimetres

Exclusion Criteria:

* Diabetes or history of other disturbances of glucose metabolism (eg impaired glucose tolerance, hypoglycaemia).
* Any genetic or psychiatric disease (e.g. fragile X syndrome, major depression) affecting brain
* Any significant chronic disease
* Renal or hepatic disease
* Recent weight changes or attempts to loose weight (> 3 kg weight gain or loss, within the last 3 months)
* Smoking (current or last 6 months)
* Alcohol consumption of more than 21 units per week or use of recreational drugs at present or in the last year
* Recent blood donation (within the last 2 months)
* Recent participation in other biomedical research projects (within the last 3 months), participation in 2 or more biomedical research projects in one year

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01-28 (Actual); Primary Completion 2013-05-23 (Actual); Study Completion 2013-05-23 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging of the hypothalamus | fMRI measurements between 8 and 20 minutes after start of beverage intake
  Hypothalamic neural activity measured using Blood Oxygen Level Dependent signal measured by functional magnetic resonance imaging

SECONDARY OUTCOMES:
Functional magnetic resonance imaging of the amygdala | fMRI measurements between 8 and 20 minutes after start of beverage intake
  Neural activity in the amygdala measured using Blood Oxygen Level Dependent signal
Functional magnetic resonance imaging of the nucleus accumbens | fMRI measurements between 8 and 20 minutes after start of beverage intake
  Neural activity in the nucleus accumbens measured using Blood Oxygen Level Dependent signal

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van der Grond, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Opstal AM, van den Berg-Huysmans AA, Hoeksma M, Blonk C, Pijl H, Rombouts SARB, van der Grond J. The effect of consumption temperature on the homeostatic and hedonic responses to glucose ingestion in the hypothalamus and the reward system. Am J Clin Nutr. 2018 Jan 1;107(1):20-25. doi: 10.1093/ajcn/nqx023. PMID 29381802